CLINICAL TRIAL: NCT04381663
Title: CSS-Assessing the Course of Degenerative Cervical Spinal Stenosis Using Functional Outcomes
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01270;ch20Muendermann
Record Dates: First submitted 2020-04-29; First posted 2020-05-11 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Cervical Spinal Stenosis; Cervical Myelopathy
Keywords: Cervical Spinal Stenosis; Cervical Myelopathy
MeSH Terms: interventions — Conservative Treatment; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- conservative treatment: In study A this group will be treated conservatively (stenosis). Study B is a single centre longitudinal study where the same patient groups will be followed up during the course of their treatment
  Interventions: Procedure: conservative treatment
- surgical treatment (stenosis and myelopathy).: In study A this group that will be treated surgically (stenosis and myelopathy). Study B is a single centre longitudinal study where the same patient groups will be followed up during the course of their treatment
  Interventions: Procedure: surgical treatment

INTERVENTIONS:
Procedure: conservative treatment — conservative treatment for patients with cervical spine stenosis without myelopathy
  Groups: conservative treatment
Procedure: surgical treatment — surgical decompress the spinal canal in patients with moderate to severe degenerative cervical spine myelopathy
  Groups: surgical treatment (stenosis and myelopathy).

SUMMARY:
The study will consist of two parts:

* In Study A, objectively assessed physical activity, gait, balance, range of movement of specific joints during walking and neurophysiological findings between patients with cervical spine stenosis (CSS) without myelopathy who will be treated conservatively and patients with stenosis and signs of myelopathy who are candidates for surgical Treatment will be compared.
* In Study B, the 6-month changes in the same outcomes in patients treated conservatively (from the first specialist consultation until 6 months later) and in patients treated surgically (preoperative day and 6-month post-operatively) will be quantified.

DETAILED DESCRIPTION:
Study A is a single centre cross-sectional study with two study groups, one that will be treated conservatively (stenosis) and one that will be treated surgically (stenosis and myelopathy).

Study B is a single centre longitudinal study where the same patient groups will be followed up during the course of their treatment.

Clinical, radiological, biomechanical (kinematic and electromyographic), neurological and neurophysiological data will be collected. Differences in and the relationship between the clinical, radiological, biomechanical, neurological and neurophysiological data will be determined .

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of degenerative cervical spine stenosis defined by MRI (stenosis grade 2 or grade 3
* Local clinical symptoms due to degenerative changes of the cervical vertebral column with or without clinically defined myelopathy

Exclusion Criteria:

* Stenosis after trauma or neoplasm
* Prior decompressive surgery
* Previous spine or extremity surgery with a consequent sensorimotor impairment
* Other pathologies than cervical spine stenosis causing gait disturbance
* BMI > 35 kg/m2
* Use of walking aids
* Inability to provide informed consent
* Contraindications for recording of Motor evoked potentials (MEP)
* Contraindications to safely undergo MRI

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with degenerative cervical spine stenosis with or without myelopathy.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Difference in gait symmetry | approximate duration: 30 minutes. Assessment will be performed at visit 1 and will be repeated 6 months after study inclusion at visit 2
  The subjects will perform an instrumented gait analysis on an overground walkway with two embedded force plates
Change in balance performance | approximate duration: 30 minutes. Assessment will be performed at visit 1 and will be repeated 6 months after study inclusion at visit 2.
  Balance performance will be assessed using the modified clinical test of sensory integration of balance (m-CTSIB) using the Biodex Balance System SD
Difference in neurophysiological outcome | approximate duration: 30 minutes. Assessment will be performed at visit 1 and will be repeated 6 months after study inclusion at visit 2.
  Quantitative score of Motor evoked potentials (MEP) and Somato-sensory evoked potentials (SEP)

SECONDARY OUTCOMES:
Difference in daily physical activity | monitored for 7 consecutive days at visit 1 or 1 week before surgery and 6 months later at visit 2
  daily physical activity will be objectively monitored for 7 consecutive days using the ActiGraph wGT3X-BT (ActiGraph Corp, Pensacola Florida, USA) worn around the hip
Difference in spinal cord gray and white matter areas | approximate duration of the scan: 30. Assessment will be performed at visit 1 and will be repeated 6 months after study inclusion at visit 2 (Measurement at visit 2 only in patients with cervical spine stenosis treated conservatively).
  Participants will be investigated on the 3 Tesla (3T) whole body MRI research scanner using 2D-Averaged Magnetization Inversion Recovery Acquisitions (AMIRA) imaging
Change in segmental quantitative muscle strength | approximate duration: 10 minutes. Assessment will be performed at visit 1 and will be repeated 6 months after study inclusion at visit 2.
  assessments of segmental muscle force via hand-held-dynamometry following the Treatment Research Initiative to Cure ALS (TRICALS) Protocol Isometric Strength Testing 2016 at each study visit
Change in 25-foot walk test | approximate duration: 3 minutes. Assessment will be performed at visit 1 and will be repeated 6 months after study inclusion at visit 2.
  time of 25-foot walk test
Change in 6-minute walk test | approximate duration: 6 minutes. Assessment will be performed at visit 1 and will be repeated 6 months after study inclusion at visit 2.
  distance of 6-minute walk test
Change in dynamic stability and range of motion during walking | approximate duration: 20 minutes. Assessment will be performed at visit 1 and will be repeated 6 months after study inclusion at visit 2.
  Subjects will first complete overground walking trials in their own shoes at normal and fast walking speed while naming months backward in a 25-m hallway while gait CSS Study Protocol Version 2, 15.8.2019 Page 12 of 21 kinematics will be recorded using the RehaGait system. Afterwards, patients will be asked to walk over the force plates in the laboratory at their preferred walking speed while kinematic, kinetic and Electromyography (EMG) data will be recorded.
Change in pain | approximate duration: 2 minutes. Assessment will be performed at visit 1 and will be repeated 6 months after study inclusion at visit 2.
  Numeric Pain Rate Scale (NPRS), a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain)
Change in function | approximate duration: 13 min. Assessment will be performed at visit 1 and will be repeated 6 months after study inclusion at visit 2
  Modified Japanese Orthopaedic Association - Scoring System (mJOA) questionnaire, This scale consists of four domain scores motor dysfunction in the upper extremities, motor dysfunction in the lower extremities, sensory function in the upper extremities and bladder function. Each scale ranges from 0 to 7, 5, 3, and 3, respectively, with a total score of 0 to 18.
  The severity of myelopathy is defined as mild if the mJOA score is 15 or larger, moderate if the mJOA score ranges from 12 to 14 or severe if the mJOA score is less than 12
Change in disability | approximate duration: 5 minutes. Assessment will be performed at visit 1 and will be repeated 6 months after study inclusion at visit 2.
  Neck Disability Index (NDI) questionnaire, a Patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation.
  The NDI has sufficient support and usefulness to retain its current status as the most commonly used self-report measure for neck pain. A score of 0-4 points means no disability, 5-14 points mild disability, 15-24 points moderate disability, 25-34 points severe disability, 35-50 points complete disability
Change in risk of falling | approximate duration: 10 minutes. Assessment will be performed at visit 1 and will be repeated 6 months after study inclusion at visit 2.
  The Berg Balance Scale (BBS) is a subjective measure for balance and risk of falling. Based on 14 items, vestibular function, balance ability, proprioception and muscle strength are assessed. The cut-off value for an elevated risk of falling is at 38 of 56 points. Older persons with a score of 45 of 56 points are able to ambulate safely and independently.

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Mündermann, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland; Cordula Netzer, Dr. med., Principal Investigator — University Hospital, Basel, Switzerland; Regina Schläger, PD Dr. med., Principal Investigator — University Hospital, Basel, Switzerland; Martin Hardmeier, PD Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Universitätsspital Basel, Basel, Switzerland